CLINICAL TRIAL: NCT04929002
Title: Using Carbon-13 Magnetic Resonance Spectroscopy to Assess Whether High Glycogen Levels in Skeletal Muscle of Patients With Glycogen Storage Diseases is a Prelude for Muscle Damage.
Brief Title: Carbon-13 Magnetic Resonance Spectroscopy in Glycogen Storage Diseases
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Research Center for Magnetic Resonance (Unknown)
Responsible Party: Principal Investigator, Mads Peter Godtfeldt Stemmerik, PhD-student, MD, Rigshospitalet, Denmark
Other Study IDs: 7TMRS in GSD
Record Dates: First submitted 2021-06-03; First posted 2021-06-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Glycogen Storage Disease; McArdle Disease; Pompe Disease (Late-onset)
MeSH Terms: conditions — Glycogen Storage Disease; Glycogen Storage Disease Type V; Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- McArdle Disease
  Interventions: Other: No intervention
- Pompe disease
  Interventions: Other: No intervention
- Controls
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The project will use carbon-13 magnetic resonance spectroscopy to assess whether high glycogen levels in skeletal muscle of patients with Glycogen Storage Diseases is a prelude for muscle damage.

Patients with Glycogen Storage Diseases will be examined using carbon-13 MR-spectroscopy to quantify the glycogen levels in lumbar, thigh and calf-muscles. The pattern of glycogen concentration will be compared to the pattern of muscle atrophy found in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with genetically verified neuromuscular disease or healthy control
* Healthy controls needs to be healthy to be included, evaluated by the investigator

Exclusion Criteria:

* Ferrous objects in or around the body
* Pacemaker or other implanted electronic devices
* Claustrophobia
* Inability to understand the purpose of the trial or corporate for the conduction of the experiments.
* Participation in other trials that may interfere with the results.
* Competing conditions at risk of compromising the results of the study, evaluated by the investigator.
* Strenuous exercise in the preceding 2 days before examination
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Pompe or McArdle disease and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Glycogen concentration | Day 1
  1. The difference in muscle glycogen between patients and controls
  2. The difference in muscle glycogen between different muscle groups in patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromuscular Research Unit, 8077, Copenhagen, Copenhange, Denmark

IPD SHARING:
Plan to Share IPD: No